CLINICAL TRIAL: NCT04628533
Title: Exploring the Optimal Duration of a Group-based Online Behavioral Weight Loss Program
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID-19. Recruitment never began.
Sponsor: University of Vermont (Other)
Collaborators: University of South Carolina (Other); University of Tennessee (Other)
Responsible Party: Principal Investigator, Jean R. Harvey, PhD, RD, Interim Dean, College of Agriculture and Life Sciences, Professor, University of Vermont
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHRBSS #STUDY00000761
Record Dates: First submitted 2020-11-02; First posted 2020-11-13 (Actual); Last update posted 2020-11-13 (Actual); Status verified 2020-11

CONDITIONS: Obesity and Overweight
MeSH Terms: conditions — Obesity; Overweight

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Four Month Duration (Experimental): Participants will meet weekly online via video chat with an experienced behavioral weight loss counselor in a synchronous 1-hour chat session for 16 weeks in a well-established behavioral weight loss program.
  Interventions: Behavioral: Four Month Duration Online Behavioral Weight Loss Program
- Six Month Duration (Active Comparator): Participants will meet weekly online via video chat with an experienced behavioral weight loss counselor in a synchronous 1-hour chat session for 24 weeks in a well-established behavioral weight loss program.
  Interventions: Behavioral: Six Month Duration Online Behavioral Weight Loss Program

INTERVENTIONS:
Behavioral: Four Month Duration Online Behavioral Weight Loss Program — Participants meet weekly on line with other group participants for 16 weeks. The group-based online behavioral weight control program incorporates the elements of current thinking and empirical data on successful weight loss programs, including restricted calorie intake and increased physical activity. Key behavioral strategies to facilitate making sustained changes in dietary habits and activity patterns are introduced, promoted, and reinforced throughout the program. Weekly "group meetings" in a video chat forum led by an experienced group weight control counselor are the venue for the group process, and extensive web-based resources to support behavior changes are offered. The online groups are "closed" such that those individuals who start the group remain in that group for the duration of their participation. Weight loss counselor will provide feedback and encouragement to participants after reviewing food diaries via weekly emails.
  Arms: Four Month Duration
Behavioral: Six Month Duration Online Behavioral Weight Loss Program — Participants meet weekly on line with other group participants for 24 weeks. The group-based online behavioral weight control program incorporates the elements of current thinking and empirical data on successful weight loss programs, including restricted calorie intake and increased physical activity. Key behavioral strategies to facilitate making sustained changes in dietary habits and activity patterns are introduced, promoted, and reinforced throughout the program. Weekly "group meetings" in a video chat forum led by an experienced group weight control counselor are the venue for the group process, and extensive web-based resources to support behavior changes are offered. The online groups are "closed" such that those individuals who start the group remain in that group for the duration of their participation. Weight loss counselor will provide feedback and encouragement to participants after reviewing food diaries via weekly emails.
  Arms: Six Month Duration

SUMMARY:
This online pilot weight loss study will explore the feasibility of recruiting individuals to an established online behavioral weight loss program of varying duration (4 months vs. 6 months), We will compare 6-month weight losses between the two programs of shorter and longer duration, respectively, and obtain data to characterize weight maintenance experiences and retention. Both groups will receive the same intervention; the only difference is the number of weeks the group will meet. Both groups will complete follow ups at 2, 4, 6, and 12 months (12 months after the study begins).

DETAILED DESCRIPTION:
Obesity presents a vexing public health challenge. Effective behavioral weight control treatments are available, loss, and projections show these interventions could have a significant impact on overall population health if the interventions were more broadly available. Internet delivery of behavioral lifestyle interventions has potential for broad reach and is thus an attractive option, although average weight losses tend to be lower than in a comparable behavioral program delivered in-person. Nonetheless, internet-delivered group behavioral weight control programs which incorporate synchronous chat "group sessions" can produce an average of 5% weight loss, with almost a quarter of participants losing at least 10% of their body weight at 6-months, and thus offer weight losses which are clinically significant. Online programs are more cost effective than in-person delivery of the same program, but efforts to optimize the delivery of online programs to achieve the best weight outcomes balanced against delivery cost are in their infancy. The current feasibility study seeks to explore critical elements to allow testing of whether a moderate dose program (16 online weekly video chat sessions) can produce weight losses comparable to the higher dose (24 weekly video chat sessions) internet-delivered behavioral weight loss program which is the established standard which we have demonstrated effective in the past. This pilot study will provide proof-of-concept to determine whether the approach is promising and if it is feasible to conduct. The pilot will explore the feasibility of recruiting individuals to weight loss programs of varying duration (4 months vs. 6 months), refine our ability to deliver the 16-session program, compare 6-month weight losses between the two programs of shorter and longer duration, respectively, and obtain data to characterize weight maintenance experiences and retention over the 12-month study period.

Up to 80 individuals will be randomized into an online behavioral weight loss program lasting 4 months or 6 months. Individuals will meet weekly for one hour in a synchronous chat session with an experienced behavioral weight control counselor. Participants will be followed over 12 months from study start.

ELIGIBILITY:
Inclusion Criteria:

* female
* BMI between 25-55
* free of medical problems that might contraindicate participation in a behavioral weight reduction program containing an exercise component
* not currently on medication that might affect weight loss
* not currently pregnant or pregnant in the previous 6 months or currently breastfeeding
* not enrolled in another weight reduction program
* must have a computer (at home or work) with access to the Internet and a video camera
* must have a smart phone (to allow use of step counting and dietary intake self-monitoring apps)
* Only one member of a household will be eligible to participate
* must successfully complete a self-monitoring diary of foods consumed for a week during screening for study eligibility
* demonstrate the ability to access the website successfully (practice chat)
* agree to be randomized to either group
* must be willing to share access to self-monitoring information collected via the app MyFitnessPal, and Fitbit.com weight data collected via the digital smart scale (scale will be provided)

Exclusion Criteria:

* have had a heart attack or a stroke in the past 6 months,
* have ever had weight loss surgery,
* have lost more than 10 pounds in the previous 6 months,
* are currently taking medications for weight loss,
* are required by their doctor to follow a special diet (other than a low fat diet)
* have plans to move from the area in the upcoming 12 months
* who have schedules that will make it likely that they will have difficulty attending the scheduled "chat" groups

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 0 (Actual)
Dates: Start 2020-07 (Estimated); Primary Completion 2021-01 (Estimated); Study Completion 2021-02 (Estimated)

PRIMARY OUTCOMES:
Change in Weight from baseline to 2, 4, 6 and 12 months | 2 months, 4 months, 6 months, 12 months
  Weight loss at each follow-up will be calculated as % kg lost from baseline.

SECONDARY OUTCOMES:
Process measures: Attendance by subjects at weekly online meetings | 2,4,6 months
  The group facilitator will take attendance at weekly online class meetings. Attendance at on-line meetings will be calculated as % of meetings actually attended out of 16 or 24 meetings that were scheduled according to condition assignment
Process measures: Completion of weekly online treatment modules by subjects | 2, 4, 6 months
  Completion of online treatment modules by each subject by condition will be calculated as % modules completed out of 16 or 24 modules scheduled according to condition assignment. Module completion is defined as viewing the module and completing the online activity questions associated with each respective module.

CONTACTS AND LOCATIONS:
Overall Officials: Jean R Harvey, PhD, Principal Investigator — University of Vermont; Delia Smith West, PhD, Principal Investigator — University of South Carolina
Locations (2):
- United States (2):
  - University of South Carolina, Columbia, South Carolina
  - Behavioral Weight Management Program/Univ of Vermont, Burlington, Vermont